CLINICAL TRIAL: NCT01399918
Title: A Phase II Trial of Everolimus and Bevacizumab in Advanced Non-Clear Cell Renal Cell Carcinoma (RCC)
Brief Title: Everolimus and Bevacizumab in Advanced Non-Clear Cell Renal Cell Carcinoma (RCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-226
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Results first posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2020-12

CONDITIONS: Renal Cell Carcinoma
Keywords: Kidney; Everolimus; Bevacizumab; 10-226; non-clear cell histology; Advanced
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Everolimus; Bevacizumab

ARMS (1):
- everolimus and bevacizumab (Experimental): This is a single-institution, single-arm phase II trial of everolimus in combination with bevacizumab in patients with advanced non-clear cell RCC, who have not received prior VEGF-.or mTOR-targeted therapy. A separate cohort of patients with non-clear cell RCC with papillary features will be enrolled in order to gather information regarding the efficacy given the rarity of these entities.
  Interventions: Drug: everolimus and bevacizumab

INTERVENTIONS:
Drug: everolimus and bevacizumab — Cycle length will be defined as 28 days. Treatment will include everolimus 10mg, self administered orally once daily on a continuous schedule (days 1-28), and bevacizumab 10mg/kg, administered intravenously on days 1 and 15 of each cycle. Treatment will be continued until disease progression, major toxicity, or withdrawal from the study for any reason. Dose modification will be permitted based on toxicity. Patients that come off study before 6 months before documented progression/death will be treated as events for the 6 month PFS endpoint.

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad the combination of two medications, everolimus and bevacizumab, has on kidney cancer. In this clinical trial we are now testing these medications in combination. We think that both together might work better that either drug alone. Importantly, both of these drugs together have been tested in patients with a different type of kidney cancer and patients tolerated the combination well.

ELIGIBILITY:
Inclusion Criteria:

* Advanced renal cell carcinoma of non-clear cell histology, histologically with papillary features confirmed by MSKCC pathology. Availability of additional tissue for correlative studies is NOT in inclusion requirement.
* Evidence of unidimensionally measurable disease per RECIST 1.1 (Eisenhauer, Therasse et al. 2009). Resolution of all acute toxic effects of prior radiotherapy or surgical procedures to NCI CTCAE Version 4.0 grade ≤1.
* Adequate organ function as defined by the following criteria:
* Absolute neutrophil count (ANC) ≥1,500/μL
* Platelets ≥100,000/μL
* Hemoglobin ≥9.0 g/dL
* Serum calcium ≤12.0 mg/dL
* Serum creatinine ≤1.5 x ULN
* Total serum bilirubin ≤2.0 x ULN
* Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) ≤2.5 x local laboratory upper limit of normal (ULN), or AST and ALT ≤5 x ULN if liver function abnormalities are due to underlying malignancy
* INR ≤1.5. (Anticoagulation is allowed if target INR ≤ 1.5 on a stable dose for >2 weeks at time of study entry.)
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.

Karnofsky performance status ≥ 70 %.

* 18 years of age or older.
* Ability to swallow oral medication.
* Signed and dated informed consent document indicating that the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to undergoing study screening procedures.
* Subject's willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Patients who have received prior systemic therapy for their RCC with VEGF pathway inhibitor (such as sunitinib, sorafenib, and bevacizumab) or with mTOR inhibitors (such as sirolimus, temsirolimus, everolimus, or deforolimus).
* Patients within 28 days post major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic), open biopsy, or significant traumatic injury to avoid wound healing complications. Minor procedures and percutaneous biopsies or placement of vascular access device without complications require 48 hours prior to study entry.
* Patients who had radiation therapy within 28 days prior to start of study treatment (palliative radiotherapy to bone lesions allowed if completed 2 weeks prior to study treatment start).

Patients with evidence or history of central nervous system (CNS) metastases or spinal cord compression, unless prior treatment with surgery or radiotherapy AND no progression of CNS disease within 6 months prior to enrollment.

* Patients with a history of abdominal fistula, gastrointestinal perforation, or intraabdominal abscess within 6 months prior to study enrollment.
* Patients with proteinuria on screening urinalysis confirmed to be >1g /24h by 24 hour urine collection.
* Patients with inadequately controlled hypertension (defined as a blood pressure of > 150 mmHg systolic and/or > 100 mmHg diastolic on medication), or any prior history of hypertensive crisis or hypertensive encephalopathy.

Patients receiving chronic systemic treatment with corticosteroids (dose of ≥ 10 mg/day methylprednisone equivalent) or another immunosuppressive agent. Inhaled and topical steroids are acceptable.

* Patients with a known history of HIV seropositivity.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * unstable angina pectoris (at any time), symptomatic congestive heart failure (NYHA III, IV) (at any time), serious uncontrolled cardiac arrhythmia (at any time), myocardial infarction, cerebrovascular accidents, or symptomatic left ventricular dysfunction ≤ 6 months prior to first study treatment
  * active bleeding diathesis
  * known severely impaired lung function defined as spirometry and DLCO ≤ 50% of normal and oxygen saturation at rest ≤ 88% on room air.
  * symptomatic intrinsic lung disease requiring oxygen supplementation at baseline
  * Uncontrolled diabetes mellitus as defined by HbA1c >8% despite adequate therapy. Patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary
  * any active (acute or chronic) or uncontrolled infection/disorders that impair the ability to evaluate the patient or for the patient to complete the study
  * liver disease such as cirrhosis decompensated liver disease or active and chronic hepatitis (i.e. quantifiable HBV-DNA and/or positive HBsAg, quantifiable HCV-RNA).
* Patients who have a history of another primary malignancy and are off treatment for ≤ 3 years, with the exception of non-melanoma skin cancer and carcinoma in situ of the uterine cervix.
* Female patients who are pregnant or breast feeding
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must use highly effective methods of contraception during the study and 8 weeks after. Highly effective contraception methods include combination of any two of the following:

  1. Use of oral, injected or implanted hormonal methods of contraception or;
  2. Placement of an intrauterine device (IUD) or intrauterine system (IUS);
  3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository;
  4. Total abstinence or;
  5. Male/female sterilization
* Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to randomization. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential.
* Male patients whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment
* Patients who are using other investigational agents or who had received investigational drugs ≤ 4 weeks prior to study treatment start.
* Patients who have received attenuated live vaccines within one week of study entry. Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines. Known intolerance or hypersensitivity to Everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus).
* Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral Everolimus.
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2011-07; Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darren Feldman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Everolimus and Bevacizumab: This is a single-institution, single-arm phase II trial of everolimus in combination with bevacizumab in patients with advanced non-clear cell RCC, who have not received prior VEGF-.or mTOR-targeted therapy.
Period: Overall Study
Arm/Group | Everolimus and Bevacizumab
Started | 57
Completed | 55
Not Completed | 2
Not completed — Not eligible and not enrolled in the study | 2

BASELINE CHARACTERISTICS:
Population: 2 participants were not eligible and were not enrolled in the study
Arm/Group | Everolimus and Bevacizumab
Number analyzed (Participants) | 55
Age, Continuous [Median (Full Range); unit: years] | 54 [19 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 44
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Efficacy of Combining Everolimus and Bevacizumab in Patients With Advanced RCC of Non-clear Cell Histology
Description: the percent of patients alive and progression-free after 6 months of therapy.
Time Frame: 6 months
Measure: Number; unit: percent of participants
Arm/Group | Everolimus and Bevacizumab
Number analyzed (Participants) | 55
percent of participants | 78

2. Secondary Outcome: Secondary Endpoint Will be the Overall Response Rate (ORR)
Description: per the international criteria defined by the Response Evaluation Criteria in Solid Tumors Committee
Time Frame: 1 year
Measure: Number; unit: percent of participants with ORR
Arm/Group | Everolimus and Bevacizumab
Number analyzed (Participants) | 55
percent of participants with ORR | 35

3. Secondary Outcome: Participants Evaluated for Toxicity
Description: Toxicity will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) v4.0 (Gompertz 1825),. Toxicities will be summarized by type and grade using frequencies and rates.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus and Bevacizumab
Number analyzed (Participants) | 55
Participants | 55

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Everolimus and Bevacizumab
All-Cause Mortality (participants affected / at risk) | 43/55
Serious Adverse Events (participants affected / at risk) | 22/55
Other Adverse Events (participants affected / at risk) | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus and Bevacizumab (N=55)
Abdominal Pain (Gastrointestinal disorders) | 6
Acute kidney injury (Renal and urinary disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Blood bilirubin increased (Investigations) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Creatinine increased (Investigations) | 5
Death NOS (General disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Fatigue (General disorders) | 2
Fever (General disorders) | 2
Flank Pain (Musculoskeletal and connective tissue disorders) | 10
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3
Hematoma (Vascular disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Lung infection (Infections and infestations) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 1
Palpitations (Cardiac disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Rectal hemorrhage (Gastrointestinal disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus and Bevacizumab (N=55)
Hypertension (Vascular disorders) | 43
Fatigue (General disorders) | 40
Mucositis oral (Gastrointestinal disorders) | 39
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 30
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 23
Nausea (Gastrointestinal disorders) | 21
Rash acneiform (Skin and subcutaneous tissue disorders) | 21
Diarrhea (Gastrointestinal disorders) | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Dry skin (Skin and subcutaneous tissue disorders) | 15
Peripheral sensory neuropathy (Nervous system disorders) | 14
Edema limbs (General disorders) | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12
Anorexia (Metabolism and nutrition disorders) | 11
Constipation (Gastrointestinal disorders) | 11
Headache (Nervous system disorders) | 10
Weight loss (Investigations) | 10
Pain (General disorders) | 9
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 8
Hypertriglyceridemia (Metabolism and nutrition disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Dysgeusia (Nervous system disorders) | 6
Urinary frequency (Renal and urinary disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 5
Alanine aminotransferase increased (Investigations) | 5
Fever (General disorders) | 5
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Alkaline phosphatase increased (Investigations) | 4
Gen disorders & admin site conditions Other, spec (General disorders) | 4
Hematuria (Renal and urinary disorders) | 4
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4
Aspartate aminotransferase increased (Investigations) | 3
Insomnia (Psychiatric disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-29): https://cdn.clinicaltrials.gov/large-docs/18/NCT01399918/Prot_SAP_000.pdf